CLINICAL TRIAL: NCT05182294
Title: Tolerance and Acute Effects of a New HFNT Nasal Cannula on Comfort, Vital Signs, Breathing Pattern and Gas Exchange in Patients Hospitalized With an Acute Exacerbation of COPD
Brief Title: Tolerance and Acute Effects of a New HFNT Nasal Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1319877
Record Dates: First submitted 2021-12-14; First posted 2022-01-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: COPD Exacerbation Acute
Keywords: Hypercapnia (PaCO2 ≥ 45 mm Hg)
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to use of the conventional symmetric nasal cannula or the new asymmetric nasal cannula and receive HFNT for 2 hours during the first session. At the end of the first session questionnaire data will be collected and ABGs will be repeated followed by a 30-minute rest period without any device. Patients will then crossover to receive HFNT via the other cannula type for another 2 hours during the second session.Inductive plethysmography will again be worn and ABGs will be obtained, and questionnaires will again be administered. At the end of this second session the patient will be discharged from the study and receive usual medical care for the COPD exacerbation and other medical conditions as clinically indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional symmetric nasal cannula (Active Comparator): The patient's breathing pattern will be assessed by inductive plethysmography while using the cannula and receive HFNT for 2 hours during the first session. Patients will then be randomized to use of the conventional symmetric nasal cannula or the new asymmetric nasal cannula. At the end of the first session questionnaire data will be collected and ABGs will be repeated followed by a 30-minute rest period without any device. Patients will then crossover to receive HFNT via the other cannula type for another 2 hours during the second session. Inductive plethysmography will again be worn and ABGs will be obtained, and questionnaires will again be administered
  Interventions: Device: AIRVO 2, the new asymmetric nasal cannula
- AIRVO 2; new asymmetric nasal cannula (Active Comparator): The patient's breathing pattern will be assessed by inductive plethysmography while using the cannula and receive HFNT for 2 hours during the first session. Patients will then be randomized to use of the conventional symmetric nasal cannula or the new asymmetric nasal cannula. At the end of the first session questionnaire data will be collected and ABGs will be repeated followed by a 30-minute rest period without any device. Patients will then crossover to receive HFNT via the other cannula type for another 2 hours during the second session. Inductive plethysmography will again be worn and ABGs will be obtained, and questionnaires will again be administered
  Interventions: Device: AIRVO 2, the new asymmetric nasal cannula

INTERVENTIONS:
Device: AIRVO 2, the new asymmetric nasal cannula — The AIRVO 2 is a humidifier with integrated flow generator that delivers warmed and humidified respiratory gases to spontaneously breathing patient through a variety of patient interfaces. This is an FDA-approved 510k device for use in hospitals and nursing homes. During HFNT, oxygen will be passed through a heated humidifier (AIRVO 2, Fisher and Paykel Healthcare) and applied continuously through conventional large-bore binasal symmetric prongs or the new asymmetric prongs cannula device, with a gas flow rate of 20-35 liters per minute or as high as the patient will tolerate and an FiO2 to keep SaO2 ≥ 90% (Airvo 2, Fisher and Paykel Healthcare). Gas flow temperature will be adjusted based on patient's comfort and range from 34-37 degrees centigrade. After completion of the study, patients will be switched back to oxygen therapy administered by nasal prongs or mask..
  Other Names: Conventional asymmetric nasal cannula

SUMMARY:
In the care of patients experiencing an acute exacerbation of COPD, supplemental oxygen therapy is often required. Oxygen is typically administered at flow rates between 1 and 4 liters per minute. High-flow nasal therapy (HFNT) has been reported to have beneficial effects in patients with hypoxemic respiratory failure and in hospitalized and non-hospitalized patients with severe COPD. Clinical efficacy in improving gas exchange depends upon patient tolerance and device-related properties such as flow rate and creation of turbulent flow in the conducting airways to improve oxygenation and carbon dioxide elimination. Alterations of nasal prong structure, such as nasal prong dimensions, may produce more robust turbulent flow at lower flow rates thereby improving gas exchange as well as patient tolerance. In this pilot study we will assess the impact of a new nasal cannula with asymmetric cannula dimensions that may create more turbulent flow at lower flow rates compared to the current symmetric nasal cannula on patient comfort as well as vital signs, pulse oximetry, breathing pattern and parameters of gas exchange in hospitalized patients with a COPD exacerbation.

DETAILED DESCRIPTION:
AIRVO 2: The AIRVO 2 is a humidifier with integrated flow generator that delivers warmed and humidified respiratory gases to spontaneously breathing patient through a variety of patient interfaces. This is an FDA-approved 510k device for use in hospitals and nursing homes. During HFNT, oxygen will be passed through a heated humidifier (AIRVO 2, Fisher and Paykel Healthcare) and applied continuously through conventional large-bore binasal symmetric prongs or the new asymmetric prongs cannula device, with a gas flow rate of 20-35 liters per minute or as high as the patient will tolerate and an FiO2 to keep SaO2 ≥ 90% (Airvo 2, Fisher and Paykel Healthcare). Gas flow temperature will be adjusted based on patient's comfort and range from 34-37 degrees centigrade. After completion of the study, patients will be switched back to oxygen therapy administered by nasal prongs or mask.

This is a pilot study in which the primary outcome is to determine the level of comfort experienced by the patient of using high-flow nasal oxygen administered by two different nasal cannulas. It is not an efficacy trial and there is no formal power analysis. All subjects are randomly assigned to two sequences, and each subject is treated subsequently with two treatments, the order of the treatments depends on its sequence. Initially, the primary endpoint and secondary endpoints will be evaluated for a carryover effect, a period effect, and a treatment effect with the use of two-tailed t-tests. We will then model treatment effects, period effects, and carryover effects using the linear mixed-effects model for this 2x2 crossover study.

Subjects may discontinue participation in the study at any point and for any reason. This decision will not be held against them in any way. If a subject decides to withdraw, the physician will assess their clinical condition and determine the best course of action for the subject. This may include alternative methods of oxygen administration. Any data that is collected up to the point of subject withdrawal will be retained for analysis.

Risks to Subjects

The AIRVO 2 is an FDA cleared device (510k number K131895). There are few expected side effects of using the AIRVO 2 device - if the humidification is too low, the subject may experience nasal/throat discomfort or epistaxis. It has been determined to be a non-significant risk device in that it meets none of the criteria for a significant risk device.

Potential Benefits to Subjects

Potential benefits of study participation include the subject experiencing a decreased work of breathing with high flow nasal therapy provided by one or both of the nasal cannulas. It is also possible that the subject will experience no direct benefit.

Privacy and Confidentiality

All data will be stored on the REDCap website. The site is 21 CFR part 11 compliant. All study personnel have been trained in human subjects protections and good clinical practices. Study data will only be accessible to study personnel via password protected websites and computer terminals.

A "HIPAA Authorization English (HRP-505)" has been provided with this submission.

Economic Burden to Subjects

All subjects will need supplemental oxygen as part of their clinical care. The only difference for this research is that the subjects will receive high-flow oxygen through two different nasal cannulas. There is no additional charge for this method of oxygen delivery.

ELIGIBILITY:
Inclusion Criteria:

i.aged ≥ 40 years (ii) hospitalization for acute exacerbation of COPD; (iii) smoker or ex-smoker (iv) FEV1 <80% of predicted and FEV1/FVC <70% postbronchodilator within 12 months prior to admission (v) have no other lung disease (including asthma) as a principal cause of pulmonary function limitation (vi) baseline PaCO2 ≥ 45 mm Hg at study entry. (vii) willing to give informed consent (viii) willing to participate in measurement of ABGs (ix) will to provide a brief history and physical examination and answer questionnaires.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Women who are known to be pregnant at the time of hospital admission
* Prisoners
* Individuals who do not understand English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Determining the level of comfort experienced by the patient of using high-flow nasal oxygen administered by two different nasal cannulas. | 6 hours
  This is a pilot study in which the primary outcome is to determine the level of comfort experienced by the patient of using high-flow nasal oxygen administered by two different nasal cannulas. The level of comfort will be assessed by a 100 mm visual analog scale from 0 (no discomfort) to 100 (maximal imaginable discomfort)
Sensation of shortness of breath | 6 hours
  Likert scale model indicating marked improvement (+2), slight improvement (+1), no change (0), slight deterioration (-1) and marked deterioration (-2) in patient's sensation of shortness of breath and overall comfort

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No